CLINICAL TRIAL: NCT00620893
Title: Bilateral, Masked Comparison of PEG-400 Based Artificial Tear vs. Systane for Dry Eye Signs, Symptoms & Refractive Regression Associated With Myopic Laser in Situ Keratomilieusis (LASIK).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Dr. Christopher Starr, Weill Cornell Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5339
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye signs and symptoms; refractive regression
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): 1. PEG-400 based artificial tear
  Interventions: Drug: PEG- 400 based artificial tear
- 2 (Active Comparator): 2. Systane
  Interventions: Drug: Systane

INTERVENTIONS:
Drug: PEG- 400 based artificial tear — Baseline: Instill one drop in the randomized eye four times daily starting the day after surgery can be used more frequently if needed Month 3: Instill one drop in the randomized eye twice daily
  Arms: 1
Drug: Systane — Baseline: Instill one drop in the randomized eye four times daily starting the day after surgery can be used more frequently if needed Month 3: Instill one drop in the randomized eye twice daily
  Arms: 2

SUMMARY:
This study will evaluate and compare 2 artificial tears in their ability to reduce post LASIK dry eye signs and symptoms. The secondary endpoint of this study is to evaluate refractive regression in these patients. The 'Refractive Outcome' data point will be defined as the difference between the post-op spherical equivalent (SE) and the pre-op targeted SE.

ELIGIBILITY:
Inclusion Criteria:

* Patients ranging from normal to mild dry eye per physician assessment
* BCVA of 20/20
* Moderate to high myopia (-3 D to -10D of sphere)
* Patients who are scheduled to under go myopic bilateral LASIK with VISX laser

Exclusion Criteria:

* Patients currently using topical cyclosporine
* Patients currently using Systane
* Patients currently using an oil-based artificial tear such as Soothe or Endura
* Any post-op epithelial defects or flap complications requiring further procedures (relifting, scraping, stretching etc.)
* DLK greater than stage 1 or infectious keratitis post-operatively
* Any uncontrolled systemic disease that may confound the results of this trial (Diabetes, Lupus, Rheumatoid Arthritis etc.)
* Anisometropia greater than 1D

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
dry eye signs | 9 months

SECONDARY OUTCOMES:
refractive regression | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Starr, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States